CLINICAL TRIAL: NCT01161017
Title: Mechanism-based Choice of Therapy for Pain: Can Successful Prevention of Migraine be Coupled to a Psychophysical Pain Modulation Profile?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Head of Neurology Department, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Migraine06CTIL
Record Dates: First submitted 2010-07-10; First posted 2010-07-13 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Migraine
Keywords: migraine patients
MeSH Terms: conditions — Migraine Disorders | interventions — Amitriptyline; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Amitriptyline. (Active Comparator): Amitriptyline
  Interventions: Drug: Amitriptyline
- 2 Topiramate (Active Comparator): Topiramate
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Amitriptyline — Initial dose of 12.5mg will be given for 2 days. Then, daily 25mg will be taken for additional 8 weeks
  Arms: 1 Amitriptyline.
Drug: Topiramate — For the first 5 days of treatment 25mg is prescribed and should be ingested in one evening dose. For another 5 days, 25g dose should be taken twice a day (morning and evening). For the next 5 days, morning dose will be 25mg; evening dose will be 50mg. For the remaining 6 weeks of treatment, a dose of 50mg twice a day will be advised
  Arms: 2 Topiramate

SUMMARY:
Mechanism-based choice of therapy for pain:

Can successful prevention of migraine be coupled to a psychophysical pain modulation profile?

ELIGIBILITY:
Inclusion Criteria:

* female and male migraine patients with a number of month attacks ≥ 4,
* age 18-75,
* without any other chronic pain.

Exclusion Criteria:

* any migraine preventive treatment for last 6 month & psychiatric,
* language or cognitive dysfunction precluding use of psychophysics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Therapeutic response to the analgesic drugs | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel